CLINICAL TRIAL: NCT07017504
Title: The Effects of a Proprioception-enhancing Assistive Orthosis on Balance and Joint Sense in Geriatric Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Science and ICT, Republic of Korea (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0720253096_1
Record Dates: First submitted 2025-05-30; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Balance; Fall Prevention; Orthotic Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proprioception-Enhancing Orthosis (Experimental): Geriatric patients with age-related diseases will undergo three assessment phases: (1) without the orthosis, (2) with the orthosis worn but vibration inactive, and (3) with the orthosis worn and vibration active.
  Interventions: Device: proprioception-enhancing assistive orthosis

INTERVENTIONS:
Device: proprioception-enhancing assistive orthosis — A wearable device that provides mechanical vibration to the tendons around the knee and ankle to enhance proprioceptive feedback. Vibration intensity and timing are controlled automatically based on body tilt measured by an IMU sensor. The device is applied during balance and joint sense assessments conducted across three visits.

SUMMARY:
This study investigates the effects of a proprioception-enhancing assistive orthosis on balance and joint sense in geriatric patients with age-related diseases. The study uses wearable devices that deliver vibration stimuli to improve proprioceptive feedback. A total of 20 participants will be enrolled in a 24-month, IRB-approved trial at Seoul National University Hospital. The study assesses functional balance and joint position sense before and after using the device.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age-related diseases affecting balance and joint sense, who meet two or more of the following criteria for sarcopenia:

   * Muscle strength: Handgrip strength < 28 kg (men), < 18 kg (women)
   * Physical performance: Short Physical Performance Battery (SPPB) ≤ 8 points
   * Muscle mass: Bioimpedance analysis showing < 7.0 kg/m² (men), < 5.7 kg/m² (women)
2. Able to fully understand and follow instructions related to walking, sitting, and balance.

Exclusion Criteria:

1. Unable or unwilling to provide informed consent
2. High risk of falls due to severe visual impairment or dizziness
3. Communication difficulties due to speech, language, or hearing problems
4. Inability to walk independently without assistive devices
5. History of diseases affecting gait, efficiency, or endurance, such as:

   * Neurological disorders (e.g., stroke, Parkinson's disease)
   * Musculoskeletal disorders affecting the lower limbs
   * History of major orthopedic surgery on the lower limbs
   * Severe back pain or musculoskeletal pain affecting gait
   * Cardiovascular disease including heart failure or uncontrolled hypertension
   * Pulmonary diseases requiring regular oxygen therapy
   * Cancer requiring treatment within the past 3 years (except for non-melanoma skin cancer or early-stage breast/prostate cancer)
   * Psychiatric disorders such as schizophrenia, other psychoses, or bipolar disorder
   * Any other disease that significantly limits mobility

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Postural Sway | up to 2 weeks
  This measures the amount of body sway during quiet standing (static) or controlled leaning in various directions (dynamic). Parameters such as center of pressure (COP) displacement, velocity, and area are recorded to assess balance stability.
  Assessments will be conducted under the following three conditions:
  1. without the orthosis,
  2. with the orthosis worn but vibration inactive, and
  3. with the orthosis worn and vibration active.

SECONDARY OUTCOMES:
Berg Balance Scale | up to 2 weeks
  The Berg Balance Scale (BBS) is a 14-item objective measure used to assess static balance and fall risk in adults. Each item is scored on a scale from 0 to 4, with 0 indicating the lowest level of function and 4 indicating the highest level. The total score ranges from 0 to 56, with higher scores indicating better balance performance.
  Assessments will be conducted under the following three conditions:
  1. without the orthosis,
  2. with the orthosis worn but vibration inactive, and
  3. with the orthosis worn and vibration active.
Romberg Test | up to 2 weeks
  The Romberg Test is a neurological test used to assess balance and proprioceptive control. Participants are asked to stand with their feet together, arms at their sides, and eyes closed, while the examiner observes for excessive sway or loss of balance. The duration for which the participant can maintain the position without stepping or falling is recorded, up to a maximum of 60 seconds. Longer durations indicate better balance.
  Assessments will be conducted under the following three conditions:
  1. without the orthosis,
  2. with the orthosis worn but vibration inactive, and
  3. with the orthosis worn and vibration active.
Passive Joint Position Reproduction Test (Passive JPR) | up to 4 weeks
  Assesses proprioceptive accuracy by passively moving a joint (e.g., the knee) to a target angle, then asking the participant to indicate when the position is reached again. The difference between target and reproduced angles reflects proprioceptive acuity.
  Assessments will be conducted under the following three conditions:
  1. without the orthosis,
  2. with the orthosis worn but vibration inactive, and
  3. with the orthosis worn and vibration active.
Active Joint Position Reproduction Test (Active JPR) | up to 4 weeks
  Participants actively move their joint to a memorized target angle without visual or auditory cues. The accuracy of the reproduced angle is used to evaluate active proprioceptive control.
  Assessments will be conducted under the following three conditions:
  1. without the orthosis,
  2. with the orthosis worn but vibration inactive, and
  3. with the orthosis worn and vibration active.
Threshold to Detection of Passive Motion (TTDPM) | up to 4 weeks
  Measures the smallest joint movement that a participant can detect while the joint is passively moved at a very slow, constant speed. This tests the sensitivity of proprioceptive input.
  Assessments will be conducted under the following three conditions:
  1. without the orthosis,
  2. with the orthosis worn but vibration inactive, and
  3. with the orthosis worn and vibration active.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno, South Korea

IPD SHARING:
Plan to Share IPD: No